CLINICAL TRIAL: NCT02623556
Title: For Tuberculosis (TB) Clinical Auxiliary Diagnosis of Recombinant Mycobacterium Tuberculosis Allergen ESAT6 - CFP10 Dose of Certain Phase III Clinical Research
Brief Title: Clinical Study of Recombinant Mycobacterium Tuberculosis ESAT6-CFP10 Allergen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: Shanghai Public Health Clinical Center (Other Government); Tianjin Haihe Hospital (Other); Air Force Military Medical University, China (Other); Proswell Medical Corporation (Industry); Wuhan Institute for Tuberculosis Control (Other); Beijing Chest Hospital (Other); Wuxi Hospital for Infectious Diseases (Other); First Affiliated Hospital of Chongqing Medical University (Other); Fuzhou Pulmonary Hospital of Fujian (Other); Zhenjiang Third People's Hospital (Unknown); Anhui Provincial Hospital (Other Government); Shenzhen Third People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: LTao-EC III-patient
Record Dates: First submitted 2015-12-03; First posted 2015-12-07 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2017-01

CONDITIONS: Tuberculosis
Keywords: diagnosis of tuberculosis; ESAT6-CFP10; skin test; diagnostic test
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TB subjects (Experimental): 720 cases TB (Tuberculosis) subjects who meet the standard respectively are divided average into two groups through a randomized and blind method.
  360 TB subjects are injected ESAT6-CFP10 (10ug/ml) in left arm and TB-PPD in right arm. 360 TB subjects are injected ESAT6-CFP10 (10ug/ml) in right arm and TB-PPD in left arm. For each of participant,the person in this clinical research, the study uniform is that every subject injects firstly left arm, observe no obvious adverse reaction, then another drug inject in right arm. Measure the induration and (or) redness of longitudinal diameter size and transverse diameter vernier caliper by vernier caliper after injection 24h, 48h and 72h.
  Interventions: Biological: ESAT6-CFP10 (10ug/ml) in left arm and TB-PPD in right arm; Biological: ESAT6-CFP10 (10ug/ml) in right arm and TB-PPD in left arm
- non-TB subjects with lung disease and suspected TB subjects (Experimental): 360 cases non-TB subjects with lung disease and suspected TB subjects,who meet the standard respectively are divided average into different groups through a randomized and blind method. 180 non-TB subjects with lung disease are injected ESAT6-CFP10(10ug/ml) in left arm and TB-PPD in right arm. 180 non-TB subjects with lung disease are injected ESAT6-CFP10 (10ug/ml) in right arm and TB-PPD in left arm. The study uniform is that every subject injects firstly left arm, observe no obvious adverse reaction, then another drug inject in right arm. Measure the induration and (or) redness of longitudinal diameter size and transverse diameter vernier caliper by vernier caliper after injection 24h, 48h and 72h.
  Interventions: Biological: ESAT6-CFP10 (10ug/ml) in left arm and TB-PPD in right arm; Biological: ESAT6-CFP10 (10ug/ml) in right arm and TB-PPD in left arm

INTERVENTIONS:
Biological: ESAT6-CFP10 (10ug/ml) in left arm and TB-PPD in right arm — All subjects including TB subjects and non-TB subjects with lung disease inject ESAT6-CFP10 (10ug/ml) in left arm and TB-PPD in right arm respectively. Two drug must use at the same participant and in different arms.
Biological: ESAT6-CFP10 (10ug/ml) in right arm and TB-PPD in left arm — All subjects including TB subjects and non-TB subjects with lung disease inject ESAT6-CFP10 (10ug/ml) in right arm and TB-PPD in left arm respectively. Two drug must use at the same participant and in different arms.

SUMMARY:
720 cases TB (Tuberculosis patients) participants、360 cases non-TB participants with lung disease and suspected TB patients who all meet the standard are divided into different groups through a randomized and blind method. Every subject inject intradermally ESAT6-CFP10 and TB-PPD (tuberculin purified protein derivative) in different arms of the same person by blind method. Specific gama-interferon (γ-IFN) detection is needed before the injection.Measure the induration and (or) redness of longitudinal diameter size and transverse diameter vernier caliper by vernier caliper after injection 24h, 48h and 72h. At the same time, we observe all kind of adverse events.

DETAILED DESCRIPTION:
Firstly, 720 cases TB (Tuberculosis) participants who meet the standard respectively are divided into different groups through a randomized and blind method.

1. ESAT6-CFP10(10ug/ml) in left arm
2. ESAT6-CFP10(10ug/ml) in right arm. Inject intradermally ESAT6-CFP10 and TB-PPD in different arms of the same participant. For each of participant, the person in this clinical research, the study uniform is that every subject injects firstly left arm, observe no obvious adverse reaction, then another drug inject in right arm. Measure the induration and (or) redness of longitudinal diameter size and transverse diameter vernier caliper by vernier caliper after injection 24h, 48h and 72h. At the same time, we observe the vital signs (breathing, heart rate, blood pressure and temperature), local reactions (rash, pain, itching and skin mucous membrane) and a variety of adverse events.

Secondly, 360 cases non-TB participants with lung disease and suspected TB participants are divided into two different groups and the procedure are as the same as 720 cases TB.

Thirdly,suspected TB participants are put under TB (Tuberculosis patients) or non-TB participants with lung disease by diagnosis when out group.

Finally, we calculate the sensitivity (positive coincidence rate) by TB (Tuberculosis patients), the specificity (negative coincidence rate) by non-TB participants with lung disease, and verify the safety and effectiveness of ESAT6-CFP10(10ug/ml) for the clinical auxiliary diagnosis of tuberculosis.

ELIGIBILITY:
Inclusion Criteria of TB (tuberculosis:include pulmonary tuberculosis and extra pulmonary tuberculosis) subjects:

* judge the pulmonary tuberculosis patient according to Health industry standard of the People's Republic of China WS288-2008:Diagnostic Criteria for pulmonary tuberculosis;
* 18 to 65 years old ,no gender limited;
* Consent and signed informed consent forms (ICF);
* Comply with follow-up.

Inclusion Criteria of extra pulmonary tuberculosis subjects:

* Diagnosed extra pulmonary tuberculosis by epidemiology, imaging, clinical symptoms, pathological examination and so on;
* Lesions outside the lungs;
* be in unfinished reinforced phase by chemotherapy;

Exclusion Criteria of TB (tuberculosis) subjects:

* Accompanied by the following severe illness:advanced cancer, diabetes, copd in acute episodes, acute/progressive liver disease or kidney disease, congestive heart failure, ect;
* Taking part in other clinical or within three months involved in any other clinical;
* Severe allergic constitution:allergic to two or more drugs;
* in pregnancy or lactation;
* in a mental illness;
* Any conditions affect the trial evaluation by investigator's judgement.

Inclusion Criteria of non-TB participants with lung disease:

* A clear lung disease but can exclude pulmonary tuberculosis by clinical symptoms, imaging, laboratory examination.
* 18 to 65 years old, no gender limited;
* Consent and signed informed consent forms (ICF);
* Comply with follow-up.

Exclusion Criteria of non-TB participants with lung disease:

* Accompanied by the following severe illness: advanced cancer, diabetes, copd in acute episodes, acute/progressive liver disease or kidney disease, congestive heart failure, ect;
* Taking part in other clinical or within three months involved in any other clinical;
* Severe allergic constitution: allergic to two or more drugs;
* in pregnancy or lactation;
* in a mental illness;
* history of tuberculosis;
* Any conditions affect the trial evaluation by investigator's judgement.

Inclusion Criteria of suspected TB participants with lung disease:

* Cases who have pulmonary tuberculosis by clinical symptoms/signs:appear cough、cough with hemoptysis、pectoralgia、dyspnea、fever（low-grade fever at afternoon）,together with night sweats、weak、loss of appetite、weight loss,and so on,or other easily-confused respiratory system disease with TB;
* 18 to 65 years old, no gender limited;
* Consent and signed informed consent forms (ICF);
* Comply with follow-up.

Exclusion Criteria of suspected TB participants with lung disease:

* Accompanied by the following severe illness: advanced cancer, diabetes, copd in acute episodes, acute/progressive liver disease or kidney disease, congestive heart failure, ect;
* Taking part in other clinical or within three months involved in any other clinical;
* Severe allergic constitution: allergic to two or more drugs;
* in pregnancy or lactation;
* in a mental illness;
* history of tuberculosis;
* Any conditions affect the trial evaluation by investigator's judgement.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1090 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Immune response of left arm (random injected ESAT6-CFP10 or PPD) from the size of induration or redness in TB patients | within 72h after injection
  We measure the size of induration or redness at 24h, 48h, 72h after administered intradermally left arm (random injected ESAT6-CFP10 or PPD)
Immune response of right arm (random injected ESAT6-CFP10 or PPD) from the size of induration or redness in TB patients | within 72h after injection
  We measure the size of induration or redness at 24h, 48h, 72h after administered intradermally right arm (random injected ESAT6-CFP10 or PPD)
Immune response of left arm (random injected ESAT6-CFP10 or PPD) from the size of induration or redness in non-TB subjects with lung disease | within 72h after injection
  We measure the size of induration or redness at 24h, 48h, 72h after administered intradermally left arm (random injected ESAT6-CFP10 or PPD)
Immune response of right arm (random injected ESAT6-CFP10 or PPD) from the size of induration or redness in non-TB subjects with lung disease | within 72h after injection
  We measure the size of induration or redness at 24h, 48h, 72h after administered intradermally right arm (random injected ESAT6-CFP10 or PPD)

SECONDARY OUTCOMES:
Number of participants with Adverse Events | within 72h after injection two drug each participant

CONTACTS AND LOCATIONS:
Overall Officials: Shuihua Lu, Bachelor, Principal Investigator — Shanghai Public Health Clinical Center; Qi Wu, Master, Principal Investigator — Tianjin Haihe Hospital; Weihua Wang, Doctor, Principal Investigator — Wuhan Institute for Tuberculosis Control; Naihui Chu, Bachelor, Principal Investigator — Beijing Chest Hospital; Qinfang Ou, Principal Investigator — Wuxi No.5 People's Hospital; Youlun Li, Doctor, Principal Investigator — First Affiliated Hospital of Chongqing Medical University; Xiaohong Chen, Principal Investigator — Fuzhou Pulmonary Hospital of fujuan; Hongqiu Pan, Principal Investigator — Zhenjiang Third People's Hospital; Xiaodong Mei, Doctor, Principal Investigator — Anhui Provincial Hospital; Qunyi Deng, Doctor, Principal Investigator — Shenzhen Third People's Hospital
Locations (2):
- China (2):
  - Wuxi NO.5 People's Hospital, Wuxi, Jiangsu
  - Shanghai Public Health clinical Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Pinxteren LA, Ravn P, Agger EM, Pollock J, Andersen P. Diagnosis of tuberculosis based on the two specific antigens ESAT-6 and CFP10. Clin Diagn Lab Immunol. 2000 Mar;7(2):155-60. doi: 10.1128/CDLI.7.2.155-160.2000. PMID 10702486
- [Background] Ravn P, Munk ME, Andersen AB, Lundgren B, Lundgren JD, Nielsen LN, Kok-Jensen A, Andersen P, Weldingh K. Prospective evaluation of a whole-blood test using Mycobacterium tuberculosis-specific antigens ESAT-6 and CFP-10 for diagnosis of active tuberculosis. Clin Diagn Lab Immunol. 2005 Apr;12(4):491-6. doi: 10.1128/CDLI.12.4.491-496.2005. PMID 15817755
- [Background] Brusasca PN, Colangeli R, Lyashchenko KP, Zhao X, Vogelstein M, Spencer JS, McMurray DN, Gennaro ML. Immunological characterization of antigens encoded by the RD1 region of the Mycobacterium tuberculosis genome. Scand J Immunol. 2001 Nov;54(5):448-52. doi: 10.1046/j.1365-3083.2001.00975.x. PMID 11696195
- [Background] Weldingh K, Andersen P. ESAT-6/CFP10 skin test predicts disease in M. tuberculosis-infected guinea pigs. PLoS One. 2008 Apr 23;3(4):e1978. doi: 10.1371/journal.pone.0001978. PMID 18431468
- [Background] Aagaard C, Govaerts M, Meikle V, Vallecillo AJ, Gutierrez-Pabello JA, Suarez-Guemes F, McNair J, Cataldi A, Espitia C, Andersen P, Pollock JM. Optimizing antigen cocktails for detection of Mycobacterium bovis in herds with different prevalences of bovine tuberculosis: ESAT6-CFP10 mixture shows optimal sensitivity and specificity. J Clin Microbiol. 2006 Dec;44(12):4326-35. doi: 10.1128/JCM.01184-06. Epub 2006 Sep 27. PMID 17005738
- See also: Center for drug evaluation, CFDA, China — http://www.cde.org.cn/
- See also: Chinese Clinical Trial Registry — http://www.chinadrugtrials.org.cn/